CLINICAL TRIAL: NCT06475443
Title: The Efficacy and Safety of Pyrotinib Plus Capecitabine in Human Epidermal Growth Factor Receptor 2-positive Breast Cancer Patients With Active Brain Metastases That Have Failed Antibody-drug Conjugate(ADC): a Prospective, Single Arm, Trial
Brief Title: Efficacy of Pyrotinib Plus Capecitabine in HER2-positive MBC With Active Brain Metastases That Have Failed ADCs
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-MBC14-BM 05
Record Dates: First submitted 2024-05-22; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Breast Cancer in the Brain
MeSH Terms: interventions — pyrotinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arms and Interventions (Experimental): HER2-positive: pyrotinib plus capecitabine
  Interventions: Drug: pyrotinib plus capecitabine

INTERVENTIONS:
Drug: pyrotinib plus capecitabine — oral
  Other Names: SHR1258

SUMMARY:
To evaluate the efficacy and safety of pyrotinib plus capecitabine in HER2-positive breast cancer patients with active brain metastases that have failed ADCs

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of pyrotinib plus capecitabine in Human Epidermal Growth Factor Receptor 2（HER2）-positive breast cancer patients with active brain metastases that have failed Antibody Drug Conjugates（Fam-trastuzumab deruxtecan-nxki[T-DXd] or A1811), had received no local radiotherapy previously and have at least one measurable brain lesion according to response assessment in neuro-oncology (RANO)criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥18 years old;
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤2;
3. Pathologically confirmed HER2-positive invasive breast cancer with metastatic disease; patients with no pathological or cytologically confirmed metastatic disease should obtain clear evidence of metastasis through physical examination or radiological examination; Note: Positive HER2 -positive refers in the pathological examination/rechecking of primary lesions or metastatic lesions performed by the Research site's Pathology Laboratory, at least once the tumour cells defined as 3+ staining by immunohistochemistry, or fluorescence in situ hybridization (FISH) confirmed positive;
4. Fam-trastuzumab deruxtecan-nxki or A1811 had failed treatment for active brain metastasis and had received no local radiotherapy previously. Patients with new lesions in the brain after craniotomy are allowed to be included, provided that radiotherapy is not performed after surgery;
5. Enhanced MRI confirmed brain metastasis. According to RANO criteria, there is at least one measurable brain lesion, and the measurability of extracranial lesions is not required;
6. Previous treatment:Capecitabine is not allowed, except for patients without progression or intolerance during use and no relapse at least 6 months (as neoadjuvant /adjuvant therapy) after discontinuation of a capecitabine-containing treatment. Pyrotinib is not allowed, except for patients without progression or intolerance during use and no relapse at least 6 months (as neoadjuvant /adjuvant therapy) after discontinuation of a pyrotinib-containing treatment ; Patients who have not previously used pyrotinib , but have used pyrotinib in the neoadjuvant / adjuvant phase, have not proven disease progression or intolerance during use, and have relapsed 6 months after the last dose are allowed to be enrolled; Concurrent use of bisphosphonates, mannitol and glucocorticoids is allowed, provided that the dosage (<2 mg dexamethasone [or equivalent])
7. Expected survival period of 3 months;
8. Patients must have adequate organ function, criteria as follows: Blood routine test (no blood transfusion within 14 days, no correction of Granulocyte colony-stimulating factor(G-CSF) and other hematopoietic stimulating factors): Absolute Neutrophil Count (ANC) 1.5X10^9 / L; PLT 75X10^9 / L; Hemoglobin（Hb） 90g / L; Blood chemistry test:total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN); Alanine transaminase(ALT) and Aspartate transaminase(AST) ≤3 times ULN; For patients with liver metastases, ALT and AST ≤5 times ULN(Upper Limit of Normal); Blood urea nitrogen(BUN) and creatinine(Cr) ≤1 times ULN and creatinine clearance ≥ 50 mL/min (CockcroftGault formula);Ultrasonic cardiogram: left ventricular ejection fraction (LVEF) ≥50%; Electrocardiograph (ECG): The QT interval corrected by Fridericia's formula (QTcF)is less than 450 ms for males and less than 470 ms for females.
9. Patients need to voluntarily join this study after they fully understand and sign the informed consent form. Patients need to have good compliance and be willing to cooperate with follow-up.

Exclusion Criteria:

1. Previous treatment for active brain metastases included other anti-tumor therapy except for T-DXd or A1811;
2. Active brain metastases requiring radiotherapy; Patients with leptomeningeal metastasis (diagnosed by imaging/positive cerebrospinal fluid cytology) or a clear indication of clinically significant leptomeningeal involvement;
3. Central Nervous System(CNS) complications that require urgent neurosurgical intervention (e.g. resection, shunt placement). Patients with poorly response brain metastases after dehydration treatment and glucocorticoid treatment, such as uncontrollable increase in intracranial pressure, jet vomiting, mental disorders, epilepsy, cognitive impairment, etc;
4. Third space fluid that cannot be controlled by drainage or other methods (such as large amounts of pleural fluid and ascites);
5. Patients who have received anti-tumor radiotherapy or surgery within 2 weeks before enrollment (minor surgery, such as tumor biopsy, thoracentesis,intravenous catheterization or the like are allowed); patients who have received endocrine therapy within 1 week before enrollment; patients who have received anti-tumor chemotherapy, molecular targeted therapy or immunotherapy before enrollment within 2 weeks or 5 half-lives from the first study dose (shorter);
6. Participated in clinical trials of other new drugs within 4 weeks before enrollment;
7. Concurrently treated, or who has been treated with HER2 tyrosine kinase inhibitors(including lapatinib, neratinib, pyrotinib, etc.);
8. History of other malignant tumours within 3 years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma , skin squamous cell carcinoma or papillary thyroid carcinoma;
9. There are serious and/or uncontrolled complications that may affect participation, including any of the following:1) Dysphagia, chronic diarrhoea and intestinal obstruction and factors that affect the administration and absorption of the drug;2) Allergic constitution; allergic to the study drug; history of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency diseases; history of organ transplantation;3) History of severe heart disease, including: myocardial infarction and heart failure; any other heart disease that is not suitable for participation (investigator assessment);4) Infection;
10. Female patients during pregnancy and lactation; fertile female patients who tested positive on a baseline pregnancy test; female patients of childbearing age who are unwilling to take effective contraceptive measures during the trial.
11. Any other circumstances that are not suitable for inclusion in this study (investigator assessment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate of Intracranial Lesion (CNS-ORR) by investigator | 2 months
  CNS-ORR was defined as percentage of participants with CNS response assessed by the investigator according to RANO-BM criteria

SECONDARY OUTCOMES:
Clinica Benifit Rate of Intracranial Lesion(CNS-CBR) by investigator | 6 months
  CNS-CBR was defined as percentage of participants with CNS response assessed by the investigator according to RANO-BM criteria
Disease Control Rate（DCR）by investigator | 6 months
  DCR was defined as percentage of participants with CNS response assessed by the investigator according to RANO-BM criteria
Progression-Free Survival (PFS) | 1.5 year
  PFS was defined as the time from first dose to first documented disease progression (PD) or death from any cause, whichever occurred first